CLINICAL TRIAL: NCT01132547
Title: Prevention of Cancer/Treatment-Related Weight Loss in Children at High Nutritional Risk
Brief Title: Cyproheptadine in Preventing Weight Loss in Children Receiving Chemotherapy for Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to slow accrual.
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SCUSF 0703; SCUSF-0703 (Other: SunCoast CCOP Research Base); 5U10CA081920-11 (NIH)
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Cancer
Keywords: cachexia; weight changes; nausea and vomiting; alveolar childhood rhabdomyosarcoma; anaplastic osteosarcoma; childhood alveolar soft-part sarcoma; childhood angiosarcoma; childhood epithelioid sarcoma; childhood fibrosarcoma; childhood gliosarcoma; childhood leiomyosarcoma; childhood liposarcoma; childhood neurofibrosarcoma; childhood synovial sarcoma; chondrosarcoma; chondrosarcomatous osteosarcoma; clear cell sarcoma of the kidney; embryonal childhood rhabdomyosarcoma; embryonal-botryoid childhood rhabdomyosarcoma; endometrial stromal sarcoma; extraosseous Ewing sarcoma; peripheral primitive neuroectodermal tumor; fibrosarcomatous osteosarcoma; localized Ewing sarcoma; localized osteosarcoma; mast cell sarcoma; metastatic childhood soft tissue sarcoma; metastatic Ewing sarcoma; metastatic osteosarcoma; mixed childhood rhabdomyosarcoma; mixed osteosarcoma; nonmetastatic childhood soft tissue sarcoma; osteoblastic osteosarcoma; ovarian carcinosarcoma; ovarian sarcoma; pleomorphic childhood rhabdomyosarcoma; previously treated childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma; recurrent adult soft tissue sarcoma; recurrent childhood gliosarcoma; recurrent childhood rhabdomyosarcoma; recurrent childhood soft tissue sarcoma; recurrent Ewing sarcoma; recurrent osteosarcoma; recurrent uterine sarcoma; small intestine leiomyosarcoma; stage I uterine sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; telangiectatic osteosarcoma; untreated childhood gliosarcoma; uterine carcinosarcoma; uterine leiomyosarcoma; localized resectable neuroblastoma; localized unresectable neuroblastoma; recurrent neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma; recurrent Wilms tumor; childhood kidney tumors; stage III Wilms tumor; stage IV Wilms tumor; childhood hepatoblastoma; childhood extracranial germ cell tumor; childhood extragonadal germ cell tumor; childhood gonadal germ cell tumor; childhood malignant ovarian germ cell tumor; childhood malignant testicular germ cell tumor; recurrent childhood malignant germ cell tumor; recurrent extragonadal germ cell tumor; recurrent extragonadal non-seminomatous germ cell tumor; recurrent malignant testicular germ cell tumor; recurrent ovarian germ cell tumor; stage III extragonadal non-seminomatous germ cell tumor; stage III malignant testicular germ cell tumor; stage IIIA ovarian germ cell tumor; stage IIIB ovarian germ cell tumor; stage IIIC ovarian germ cell tumor; stage IV extragonadal non-seminomatous germ cell tumor; stage IV ovarian germ cell tumor; recurrent childhood medulloblastoma; untreated childhood medulloblastoma; childhood ependymoblastoma; childhood infratentorial ependymoma; newly diagnosed childhood ependymoma; recurrent childhood ependymoma; recurrent childhood subependymal giant cell astrocytoma; untreated childhood subependymal giant cell astrocytoma; peripheral primitive neuroectodermal tumor of the kidney; childhood supratentorial primitive neuroectodermal tumor; recurrent childhood brain stem glioma; recurrent childhood brain tumor; untreated childhood brain stem glioma; recurrent childhood anaplastic astrocytoma; recurrent childhood anaplastic oligoastrocytoma; recurrent childhood anaplastic oligodendroglioma; stage I childhood anaplastic large cell lymphoma; stage II childhood anaplastic large cell lymphoma; stage III childhood anaplastic large cell lymphoma; stage IV childhood anaplastic large cell lymphoma; untreated childhood anaplastic astrocytoma; untreated childhood anaplastic oligoastrocytoma; untreated childhood anaplastic oligodendroglioma; childhood high-grade cerebellar astrocytoma; childhood low-grade cerebellar astrocytoma; recurrent childhood astrocytoma; other tumor of glial origin; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood diffuse astrocytoma; recurrent childhood fibrillary astrocytoma; recurrent childhood gemistocytic astrocytoma; recurrent childhood oligoastrocytoma; recurrent childhood pilocytic astrocytoma; recurrent childhood pilomyxoid astrocytoma; recurrent childhood pleomorphic xanthoastrocytoma; recurrent childhood protoplasmic astrocytoma; untreated childhood cerebellar astrocytoma; untreated childhood cerebral astrocytoma; untreated childhood diffuse astrocytoma; untreated childhood fibrillary astrocytoma; untreated childhood gemistocytic astrocytoma; untreated childhood oligoastrocytoma; untreated childhood pilocytic astrocytoma; untreated childhood pilomyxoid astrocytoma; untreated childhood pleomorphic xanthoastrocytoma; untreated childhood protoplasmic astrocytoma; recurrent childhood gliomatosis cerebri; recurrent childhood oligodendroglioma; recurrent childhood visual pathway; hypothalamic glioma; recurrent childhood visual pathway glioma; untreated childhood gliomatosis cerebri; untreated childhood oligodendroglioma; untreated childhood visual pathway; untreated childhood visual pathway glioma; recurrent childhood giant cell glioblastoma; recurrent childhood glioblastoma; untreated childhood giant cell glioblastoma; untreated childhood glioblastoma; childhood choroid plexus tumor; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; minimally differentiated myeloid leukemia (M0); myeloblastic leukemia with maturation (M2); myeloblastic leukemia without maturation (M1); childhood acute myelomonocytic leukemia (M4); childhood acute promyelocytic leukemia (M3); recurrent childhood acute myeloid leukemia; untreated childhood acute myeloid leukemia; other myeloid malignancies; childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); unspecified childhood solid tumor
MeSH Terms: conditions — Neoplasms; Cachexia; Body Weight Changes; Nausea; Vomiting; Hemangiosarcoma; Sarcoma; Fibrosarcoma; Liposarcoma; Chondrosarcoma; Sarcoma, Endometrial Stromal; Neuroectodermal Tumors, Primitive, Peripheral; Mast-Cell Sarcoma; Sarcoma, Ewing; Osteosarcoma; Bone Neoplasms; Neuroblastoma; Wilms Tumor; Hepatoblastoma; Ovarian Germ Cell Cancer; Testicular Neoplasms; Medulloblastoma; Familial ependymoma; Astrocytoma; Oligodendroglioma; Lymphoma, Large-Cell, Anaplastic; Neoplasms, Neuroepithelial; Optic Nerve Glioma; Glioblastoma; Choroid Plexus Neoplasms | interventions — Cyproheptadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I cyproheptadine hydrochloride (Experimental): Patients receive oral cyproheptadine hydrochloride twice daily for 8 weeks.
  Interventions: Drug: cyproheptadine hydrochloride
- Arm II placebo (Placebo Comparator): Patients receive an oral placebo twice daily for 8 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: cyproheptadine hydrochloride — Given orally
  Other Names: cyproheptadine HCl
  Arms: Arm I cyproheptadine hydrochloride
Other: placebo — Given orally
  Arms: Arm II placebo

SUMMARY:
RATIONALE: Cyproheptadine hydrochloride may prevent weight loss caused by cancer or cancer treatment. It is not yet known whether cyproheptadine is more effective than a placebo in preventing weight loss in young patients receiving chemotherapy for cancer.

PURPOSE: This randomized phase III trial is studying cyproheptadine hydrochloride to see how well it works in preventing weight loss in young patients receiving chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the effect of cyproheptadine hydrochloride in the prevention of cancer- or treatment-related weight loss (defined as ≥ 5% reduction in weight from baseline measurement) in children who are initiating a course of moderately or highly emetic chemotherapy.

Secondary

* To investigate the effect of cyproheptadine HCl on the change in weight for age scores after 8 weeks of study drug administration in comparison to placebo.
* Investigate the relationship between the secondary outcome variables (prealbumin, triceps skin fold, mid-upper arm circumference, and weight loss)from baseline to end of treatment in each group (treatment and placebo) separately.

OUTLINE: This is a multicenter study. Patients are stratified according to enrolling center and steroid use with cancer treatment (yes vs no). Study agent can start anytime up to and including day 28 after the first dose of chemotherapy.

* Arm I: Patients receive oral cyproheptadine hydrochloride twice daily for 8 weeks.
* Arm II: Patients receive an oral placebo twice daily for 8 weeks.

Patients undergo weight and height measurements at baseline and at each follow-up visit in weeks 4 and 8 to evaluate the effect of cyproheptadine hydrochloride and duration of response. Patients or parents complete medicine logs at each follow-up visit in weeks 4 and 8 to evaluate drug compliance and tolerance. Patients also undergo measures of nutrition; and measures of body composition, lean body mass, and fat percentage using standardized equipment and procedures for measuring triceps skin fold and mid-arm muscle circumference at baseline and at the end of the study.

Patients undergo blood sample collection at baseline and at the end of the study for biomarker studies. Samples are analyzed for pre-albumin levels.

ELIGIBILITY:
INCLUSION CRITERIA:

* ≥ 2 years and ≤ 21 years of age at the time of study entry
* Scheduled to receive chemotherapy for:
* Newly diagnosed:
* Non-rhabdo soft tissue sarcomas, scheduled to receive chemotherapy, as well as intermediate or high-risk rhabdomyosarcoma, any stage osteosarcoma and any stage Ewing's sarcoma
* Intermediate or high-risk neuroblastoma
* Wilms' tumor (Stage III/IV)
* Hepatoblastoma (Stage III/IV)
* Germ cell tumors (Stage III/IV)
* Brain tumors, including medulloblastoma, PNET and ependymomas
* AML
* Relapsed/recurrent disease (any patient)
* Able to register and randomize within 28 days of starting chemotherapy (registration /randomization and start of study agent may occur at anytime up to and including Day 28 after the initiation of chemotherapy)

EXCLUSION CRITERIA:

* ≥ 29 days after starting chemotherapy
* Documented history of unintended weight loss ≥ 5% presumed secondary to cancer within 3 months of study entry
* Currently taking cyproheptadine HCl (or have taken cyproheptadine HCl within 3 weeks of study registration)
* History of anorexia nervosa or bulimia
* Taking other appetite-stimulating medications, i.e. dronabinol (Marinol) during the past three weeks.
* Initiation of other appetite enhancing agents, including steroids prescribed for the intent of weight gain, i.e. Megace. Note: Other forms of nutrition therapies, e.g. appetite-stimulating medications, TPN or enteral tube feedings are not allowed during this study.
* Children receiving steroids for >7 days as part of their cancer treatment regimen are excluded from participation. However, intermittent steroid use in an antiemetic regimen is allowed during the study
* Receiving monoamine oxidase (MAO) inhibitors, procarbazine, fluoxetine (Prozac), or paroxetine (Paxil)
* Diagnosed with glaucoma, cystic fibrosis, inflammatory bowel disease, or GI/GU obstruction
* Allergy to cyproheptadine HCl
* Females of childbearing age must not be pregnant.
* Female patients who are lactating must agree to stop breast-feeding.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2010-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey P. Krischer, PhD, Principal Investigator — University of South Florida
Locations (14):
- United States (14):
  - Miller Children's Hospital, Long Beach, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - A.I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Southwest Florida at Lee Memorial, Fort Myers, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Hospital Pensacola, Pensacola, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Columbia University Medical Center, New York, New York
  - CHRISTUS Santa Rosa Children's Hospital, San Antonio, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I Cyproheptadine Hydrochloride | Arm II Placebo
Started | 9 | 13
Completed | 5 | 12
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I Cyproheptadine Hydrochloride | Arm II Placebo | Total
Number analyzed (Participants) | 9 | 13 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (5.7) | 12.0 (4.7) | 11.2 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Participant With Weight Loss ≥ 5% at the 8- Week Assessment When Compared to Baseline
Time Frame: 8 weeks
Population: LOCF
Measure: Number; unit: participants
Arm/Group | Arm I Cyproheptadine Hydrochloride | Arm II Placebo
Number analyzed (Participants) | 9 | 13
participants | 0 | 2

2. Primary Outcome: Severity of Weight Loss
Description: Change from Baseline in Weight Z score
Time Frame: Baseline and 8 weeks
Population: Completers =
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Arm I Cyproheptadine Hydrochloride | Arm II Placebo
Number analyzed (Participants) | 5 | 12
Z score | 0.12 (1.15) | -0.02 (0.30)

3. Secondary Outcome: Pattern of Weight in the Study Population
Description: Change from Baseline in Weight
Time Frame: Baseline and 8 weeks
Population: Completers
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Arm I Cyproheptadine Hydrochloride | Arm II Placebo
Number analyzed (Participants) | 5 | 12
Kilograms | 0.18 (0.79) | -0.32 (3.13)

ADVERSE EVENTS:
Arm/Group | Arm I Cyproheptadine Hydrochloride | Arm II Placebo
Serious Adverse Events (participants affected / at risk) | 3/9 | 0/13
Other Adverse Events (participants affected / at risk) | 4/9 | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I Cyproheptadine Hydrochloride (N=9) | Arm II Placebo (N=13)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decrease (Investigations) | 2 (2) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Neutrophil count decrease (Investigations) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I Cyproheptadine Hydrochloride (N=9) | Arm II Placebo (N=13)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Skin and Subcutaneous tissue disorders other (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Tachycardia NOS (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes